CLINICAL TRIAL: NCT05613673
Title: Comparison of the Prognostic Value of Different Nutritional Assessment Scores Regarding the Course in Acute Pancreatitis - a Prospective Trial
Brief Title: Prognostic Value of Different Nutritional Screening Tools in Acute Pancreatitis
Acronym: NuRiPa
Status: Active, not recruiting | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 112/22
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Pancreatitis; Malnutrition
Keywords: Acute pancreatitis; Nutritional screening
MeSH Terms: conditions — Pancreatitis; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - observational study only — No intervention - observational study only

SUMMARY:
The goal of this observational study is to compare the prognostic value of different nutritional screening tools to predict the course of acute pancreatitis.

The main questions it aims to answer are:

* Which nutritional screening tool performs best to predict length of hospital stay?
* Which nutritional screening tool performs best to predict clinical outcome (disease severity, length of hospital stay, mortality, need for rehospitalization)?

Participants will answer questions regarding their nutritional status and undergo basic anthropometric assessments (e.g. measurement of waist circumference) to evaluate their risk of malnutrition.

DETAILED DESCRIPTION:
Malnutrition seems to be related to an adverse outcome of acute pancreatitis. However, it is still unclear which of the various available nutritional screening tools is suited best to predict the clinical outcome in hospitalized patients with acute pancreatitis.

Therefore, in this study we compare the predictive performance of 6 different nutritional screening tools that are commonly applied in clinical practice regarding their respective associations with severity of acute pancreatitis, length of hospital stay, mortality and need for rehospitalization.

To determine patients' nutritional status, subjects will be inquired about their recent food intake as well as body weight and undergo basic anthropometric assessments according to the different screening tools.

Six months after the initial diagnosis patients will be contacted via mail to report on need for rehospitalization due to acute pancreatitis during this time period.

ELIGIBILITY:
Inclusion Criteria:

* verified diagnosis of acute pancreatitis
* provision of informed consent

Exclusion Criteria:

* pregnancy
* inability to provide consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at University Medicine Greifswald (Northeast Germany). Patients admitted to the hospital for treatment of acute pancreatitis will be identified in the respective wards and will be approached for study inclusion upon confirmation of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Relation of Nutritional Risk Screening 2002 to length of hospital stay | Baseline
  Association between Nutritional Risk Screening 2002 (NRS-2002) result and length of hospital stay. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.

SECONDARY OUTCOMES:
Relation of Nutritional Risk Index to length of hospital stay | Baseline
  Association between Nutritional Risk Index (NRI) result and length of hospital stay. NRI is a continuous measure, with lower values indicating greater nutritional risk.
Relation of Mini Nutritional Assessment - Short Form to length of hospital stay | Baseline
  Association between Mini Nutritional Assessment - Short Form (MNA-SF) result and length of hospital stay. MNA-SF score ranges from 0 to 14, with lower values indicating greater nutritional risk.
Relation of Subjective Global Assessment to length of hospital stay | Baseline
  Association between Subjective Global Assessment result and length of hospital stay. SGA scores of A, B, and C indicate no malnutrition, moderate malnutrition or severe malnutrition, respectively.
Relation of Malnutrition Universal Screening Tool to length of hospital stay | Baseline
  Association between Malnutrition Universal Screening Tool (MUST) result and length of hospital stay. MUST score ranges from 0 to 6, with higher values indicating greater nutritional risk.
Relation of Short Nutritional Assessment Questionaire to length of hospital stay | Baseline
  Association between Short Nutritional Assessment Questionaire (SNAQ) result and length of hospital stay. SNAQ score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of fat-free mass to length of hospital stay | Baseline
  Association between fat-free mass determined by bioelectrical impedance analysis and length of hospital stay.
Relation of fat mass to length of hospital stay | Baseline
  Association between fat mass determined by bioelectrical impedance analysis and length of hospital stay.
Relation of skeletal muscle mass to length of hospital stay | Baseline
  Association between skeletal muscle mass determined by computed tomography and length of hospital stay.
Relation of waist circumference to length of hospital stay | Baseline
  Association between waist circumference and length of hospital stay.
Relation of albumin to length of hospital stay | Baseline
  Association between plasma albumin concentration at admission and length of hospital stay.
Relation of C-reactive protein to length of hospital stay | Baseline
  Association between plasma C-reactive protein concentration at admission and length of hospital stay.
Relation of Nutritional Risk Screening 2002 to disease severity | Baseline
  Association between Nutritional Risk Screening 2002 (NRS-2002) result and severity of acute pancreatitis based on the Revised Atlanta Classification. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Nutritional Risk Index to disease severity | Baseline
  Association between Nutritional Risk Index (NRI) result and severity of acute pancreatitis based on the Revised Atlanta Classification. NRI is a continuous measure, with lower values indicating greater nutritional risk. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Mini Nutritional Assessment - Short Form to disease severity | Baseline
  Association between Mini Nutritional Assessment - Short Form (MNA-SF) result and severity of acute pancreatitis based on the Revised Atlanta Classification. MNA-SF score ranges from 0 to 14, with lower values indicating greater nutritional risk. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Subjective Global Assessment to disease severity | Baseline
  Association between Subjective Global Assessment (SGA) result and severity of acute pancreatitis based on the Revised Atlanta Classification. SGA scores of A, B, and C indicate no malnutrition, moderate malnutrition or severe malnutrition, respectively. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Malnutrition Universal Screening Tool to disease severity | Baseline
  Association between Malnutrition Universal Screening Tool (MUST) result and severity of acute pancreatitis based on the Revised Atlanta Classification. MUST score ranges from 0 to 6, with higher values indicating greater nutritional risk. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Short Nutritional Assessment Questionaire to disease severity | Baseline
  Association between Short Nutritional Assessment Questionaire (SNAQ) result and severity of acute pancreatitis based on the Revised Atlanta Classification. SNAQ score ranges from 0 to 7, with higher values indicating greater nutritional risk. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of fat-free mass to disease severity | Baseline
  Association between fat-free mass determined by bioelectrical impedance analysis and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of fat mass to disease severity | Baseline
  Association between fat mass determined by bioelectrical impedance analysis and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of skeletal muscle mass to disease severity | Baseline
  Association between skeletal muscle mass determined by computed tomography and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of waist circumference to disease severity | Baseline
  Association between waist circumference and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of albumin to disease severity | Baseline
  Association between plasma albumin concentration at admission and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of C-reactive protein to disease severity | Baseline
  Association between plasma C-reactive protein concentration at admission and severity of acute pancreatitis based on the Revised Atlanta Classification. Based on the Revised Atlanta Classification acute pancreatitis can be graded as mild, moderate, or severe.
Relation of Nutritional Risk Screening 2002 to mortality | Baseline
  Association between Nutritional Risk Screening 2002 (NRS-2002) result and in-hospital mortality. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of Nutritional Risk Index to mortality | Baseline
  Association between Nutritional Risk Index (Index) result and in-hospital mortality. NRI is a continuous measure, with lower values indicating greater nutritional risk.
Relation of Mini Nutritional Assessment - Short Form to mortality | Baseline
  Association between Mini Nutritional Assessment - Short Form (MNA-SF) result and in-hospital mortality. MNA-SF score ranges from 0 to 14, with lower values indicating greater nutritional risk.
Relation of Subjective Global Assessment to mortality | Baseline
  Association between Subjective Global Assessment (SGA) result and in-hospital mortality. SGA scores of A, B, and C indicate no malnutrition, moderate malnutrition or severe malnutrition, respectively.
Relation of Malnutrition Universal Screening Tool to mortality | Baseline
  Association between Malnutrition Universal Screening Tool (MUST) result and in-hospital mortality. MUST score ranges from 0 to 6, with higher values indicating greater nutritional risk.
Relation of Short Nutritional Assessment Questionaire to mortality | Baseline
  Association between Short Nutritional Assessment Questionaire (SNAQ) result and in-hospital mortality. SNAQ score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of fat-free mass to mortality | Baseline
  Association between fat-free mass determined by bioelectrical impedance analysis and in-hospital mortality.
Relation of fat mass to mortality | Baseline
  Association between fat mass determined by bioelectrical impedance analysis and in-hospital mortality.
Relation of skeletal muscle mass to mortality | Baseline
  Association between skeletal muscle mass determined by computed tomography and in-hospital mortality.
Relation of waist circumference to mortality | Baseline
  Association between waist circumference and in-hospital mortality.
Relation of albumin to mortality | Baseline
  Association between plasma albumin concentration at admission and in-hospital mortality.
Relation of C-reactive protein to mortality | Baseline
  Association between plasma C-reactive protein concentration at admission and in-hospital mortality.
Relation of Nutritional Risk Screening 2002 to rehospitalization | 6 months after initial hospital admission
  Association between Nutritional Risk Screening 2002 (NRS-2002) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. NRS-2002 score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of Nutritional Risk Index to rehospitalization | 6 months after initial hospital admission
  Association between Nutritional Risk Index (NRI) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. NRI is a continuous measure, with lower values indicating greater nutritional risk.
Relation of Mini Nutritional Assessment - Short Form to rehospitalization | 6 months after initial hospital admission
  Association between Mini Nutritional Assessment - Short Form (MNA-SF) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. MNA-SF score ranges from 0 to 14, with lower values indicating greater nutritional risk.
Relation of Subjective Global Assessment to rehospitalization | 6 months after initial hospital admission
  Association between Subjective Global Assessment (SGA) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. SGA scores of A, B, and C indicate no malnutrition, moderate malnutrition or severe malnutrition, respectively.
Relation of Malnutrition Universal Screening Tool to rehospitalization | 6 months after initial hospital admission
  Association between Malnutrition Universal Screening Tool (MUST) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. MUST score ranges from 0 to 6, with higher values indicating greater nutritional risk.
Relation of Short Nutritional Assessment Questionaire to rehospitalization | 6 months after initial hospital admission
  Association between Short Nutritional Assessment Questionaire (SNAQ) result and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital. SNAQ score ranges from 0 to 7, with higher values indicating greater nutritional risk.
Relation of fat-free mass to rehospitalization | 6 months after initial hospital admission
  Association between fat-free mass determined by bioelectrical impedance analysis and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.
Relation of fat mass to rehospitalization | 6 months after initial hospital admission
  Association between fat mass determined by bioelectrical impedance analysis and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.
Relation of skeletal muscle mass to rehospitalization | 6 months after initial hospital admission
  Association between skeletal muscle mass determined by computed tomography and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.
Relation of waist circumference to rehospitalization | 6 months after initial hospital admission
  Association between waist circumference and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.
Relation of albumin to rehospitalization | 6 months after initial hospital admission
  Association between plasma albumin concentration at admission and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.
Relation of C-reactive protein to rehospitalization | 6 months after initial hospital admission
  Association between plasma C-reactive protein concentration at admission and number of rehospitalizations due to acute pancreatitis within 6 months after initial admission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Aghdassi, Professor, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany